CLINICAL TRIAL: NCT06276413
Title: Registry on Gore Branch Endoprosthesis
Brief Title: REgistRy BRAnch goRE EndopRosthEsis
Acronym: REBRA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Michele Piazza, MD, University Hospital Padova
Other Study IDs: REBRA; REBRA (Registry Identifier: REBRA)
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Aortic Aneurysm, Thoracic; Aortic Dissection
Keywords: endograft
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: GORE TAG Thoracic Branch Endoprosthesis — deployment of the GORE TAG Thoracic Branch Endoprosthesis fro thoraci aorta pathologies

SUMMARY:
Multicenter registry on patients treated by the new Gore thoracic branched endoprosthesis

DETAILED DESCRIPTION:
This is a multicenter, non-sponsored, physician-initiated multicenter registry on patients treated with the Gore thoracic branched endoprosthesis.

Inclusion of centers is on a voluntary basis; each participating center includes consecutive patients treated with this device.

ELIGIBILITY:
Inclusion Criteria:

* patients receving the Gore TAG thoracic branched endograft for thoracic aorta pathologies

Exclusion Criteria:

* less than 18 years
* allergy to endograft components
* patients receiving other types of arch endografts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated with the Gore TAG thoracic branched endograft in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
early mortality | 30 days
  mortality related to the intervention within 30 days
device stability | 5 years
  freedom from related mortality, reintervention, type 1a endoleak during follow-up
technical success | 30 days
  succesful deployment of all endograft components at the intended site with complete aneurysm exclusion, without surgical conversion, type Ia/III endoleak, kink, stenosis, graft occlusion

SECONDARY OUTCOMES:
early major adverse events | 30 days
  stroke, spinal cord ischemia, vascular complications, cardiac complications, respiratory insufficiency, early reintervention, acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular and Endovascular Clinic - Padova University, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided